CLINICAL TRIAL: NCT04970121
Title: A Single-Center, Single-Arm Clinical Trail Evaluating Efficacy and Safety of Duloxetine in Chinese Solid Tumor Patients with Taxanes-induced Painful Peripheral Neuropathy
Brief Title: Efficacy and Safety of Duloxetine in Chinese Solid Tumor Patients with Taxanes-induced Painful Peripheral Neuropathy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yan Yang, MD, Ph.D (Other)
Responsible Party: Sponsor-Investigator, Yan Yang, MD, Ph.D, Associate Director of the Department of Medical Oncology, The First Affiliated Hospital of Bengbu Medical University
Organization: The First Affiliated Hospital of Bengbu Medical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BYEC20210701
Record Dates: First submitted 2021-07-16; First posted 2021-07-21 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy; Pain; Solid Tumor
Keywords: Chemotherapy-induced Peripheral Neuropathy; Pain; Duloxetine; Taxanes; Solid tumor
MeSH Terms: conditions — Pain | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Intervention Model Description: Duloxetine treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Duloxetine arm (Experimental): Chemotherapy regimens consisting of taxanes will be used according to treatment specifications. Subjects require therapeutic intervention for painful peripheral neuropathy will receive duloxetine 20 mg (orally, once daily) as the starting dose for 1 cycle of 7 days; the current dose will be maintained for effective pain control (NRS ≤ 3 points) and increased by 20 mg at the next cycle assessment for ineffective pain control (NRS > 3 points) up to a maximum dose of 60 mg (orally, once daily). Duloxetine administration will be maintained until the uncontrolled pain (under the condition of treatment with duloxetine at its maximum dose), intolerable toxicity, completed antineoplastic therapy or subject loss of visit, death, withdrawal of informed consent, or other conditions occur. The administration of duloxetine is up to a maximum of 12 weeks.
  Interventions: Drug: Duloxetine

INTERVENTIONS:
Drug: Duloxetine — Duloxetine, tablets, 20mg as starting dose and up to 60mg as maximum dose, once daily.
  Taxanes is used according to manual instruction and patient condition.
  Other Names: Chemotherapy containing taxanes

SUMMARY:
The study is to evaluate the efficacy and safety of duloxetine in Chinese solid tumor patients with taxanes-induced painful peripheral neuropathy. Duloxetine will be given to patients who have grade 1 or higher sensory neuropathy according to the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 and at least 4 on a scale of 0 to 10 points, representing average chemotherapy-induced pain, after taxanes treatment. Patient-reported pain severity, functional interference, emotion condition and quality of Life will be assessed weekly using corresponding scales. Blood samples will be collected from each enrolled subjects before the start of treatment, and the potential biomarkers in predicting duloxetine efficacy or safety will be explored by genomic profiling.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must sign an informed consent form (ICF) voluntarily and be able to understand and comply with the requirements of the study;
2. Patients must be 18 to 75 years of age (including cut-offs) on the date of signing the informed consent form, regardless of gender;
3. Patients must be diagnosed with malignant solid tumors by pathological histology or cytology in the central laboratory or study center;
4. Patients must received treatment with a chemotherapy regimen containing taxanes;
5. Patients must have ≥ grade 1 sensory chemotherapy-induced peripheral neuropathy (CIPN) with NRS ≥ 4/10 according to the NCI Common Toxicity Criteria for Adverse Events (CTCAE) v.5.0 grading scale
6. Eastern Cooperative Oncology Group performance status (ECOG PS): 0-2;
7. Expected survival of ≥ 3 months;
8. Screening values at screening meet the following requirements: (no blood components, cell growth factors, leukocyte-lifting drugs, platelet-lifting drugs, anemia-correcting drugs, etc. are allowed within 14 days prior to obtaining laboratory tests); Complete blood count: neutrophil count (ANC) ≥ 1.5 × 109/L, platelet count (PLT) ≥ 90 × 109/L, hemoglobin (Hb) ≥ 90 g/L; Liver function: glutamic aminotransferase (AST), alanine aminotransferase (ALT) and total serum bilirubin (TBIL) ≤ 2 times the upper limit of normal range (ULN) Renal function: serum creatinine (Cr) ≤ ULN or creatinine clearance (CCr) ≥ 80 mL/min (applying the standard Cockcroft -Gault formula);
9. Female patients who are non-lactating and must have a negative pregnancy test result;
10. Patients of childbearing potential must agree to use effective contraception for at least 30 days after signing the informed consent to the last dose.

Note: Concomitant use of selected analgesics (e.g., opioids, acetaminophen, aspirin, and other NSAIDs) is permitted, but only patients receiving a stable dose during the two weeks prior to enrollment may participate.

Exclusion Criteria:

1. Patients with known hypersensitivity to duloxetine or any of the inactive ingredients in the product;
2. Patients on other concomitant medications known to affect 5-hydroxytryptamine (5-HT) levels;
3. Patients who must take monoamine oxidase inhibitors for antidepressant treatment；
4. Patients with the presence of active brain or meningeal metastases；
5. Patients with the presence of uncontrolled closed-angle glaucoma；
6. Patients with the presence of neuropathy caused by any type of nerve compression；
7. The presence of mental illness, epilepsy, mania, suicidal depression, dementia or alcohol or drug abuse that may have an impact on compliance with trial requirements;
8. The presence of comorbid cardiovascular disease, including but not limited to: (1) New York Heart Association (NYHA) criteria ≥ grade 2 heart failure; (2) severe/unstable angina pectoris; (3) myocardial infarction or cerebrovascular accident within 6 months prior to first dose; (4) atrial fibrillation and supraventricular or ventricular arrhythmias requiring treatment; (5) pre-existing symptomatic superior vena cava syndrome; (6) corrected QT interval (QTc) > 450 ms (men); QTc > 470 ms (women); (7) hypertensive disease not controlled by antihypertensive medication: systolic blood pressure ≥ 140 mmHg or diastolic blood pressure ≥ 90 mmHg;
9. Patients with other medical history or evidence of disease that has the potential to confound trial results are excluded from the study；
10. Patients are excluded from the study if investigator/sponsor believes that participation in the study is not in the subject's best interest.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-08-21 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Pain Score | Once every 7 days after treatment initiation.
  Scale title: Brief Pain Inventory Short Form (BPI-SF). Description: Pain severity items are scored using an 11-point numeric rating scale (0, no pain; 10, pain as bad as you can imagine).

SECONDARY OUTCOMES:
Quality of Life Score | Once every 7 days after treatment initiation.
  Scale title: Functional Assessment of Cancer Therapy/Gynecologic Oncology Group-Neurotoxicity (FACT/GOG-Ntx) Description: Items in FACT/GOG-Ntx are scored using an 5-point numeric rating scale (0, not at all; 4, very much).
Function Score | Once every 7 days after treatment initiation.
  Scale title: Brief Pain Inventory Short Form (BPI-SF). Description: Degree of pain-related functional interference is based on partial items in the BPI-SF and scored using an 11-point numeric rating scale, (0, does not interfere; 10, completely interferes).
Anxiety and depression Score | Once every 7 days after treatment initiation.
  Scale 1 title: Hamilton Anxiety Rating Scale (HAM-A) Description: Each item is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-56, where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe.
  Scale 2 title: Hamilton Depression Rating Scale (HDRS17) Description: HDRS17 uses a 5-point scale of 0 to 4 for most items and a 3-point scale of 0 to 2 for a few items, and higher scores mean a worse symptom. The total scores less than 7 or 7 are indicative of the absence of depression or being normal, 8-16 consider mild depression, 17-23 suggest moderate depression and scores 24 or over are indicative of severe depression.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Yang, M.D.,Ph.D, Principal Investigator — First Affiliated Hospital of Bengbu Medical College
Locations (1):
- Jing Liu, Bengbu, Anhui, China

IPD SHARING:
Plan to Share IPD: No